CLINICAL TRIAL: NCT04087551
Title: Incidence of Near-falls and the Development of the Balance Recovery Falls-efficacy Scale (BRFES) for the Community-dwelling Older Adults.
Brief Title: Development of the Balance Recovery Falls-Efficacy Scale for the Community-dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Margaret University (Other)
Collaborators: Singapore Institute of Technology (Other)
Responsible Party: Principal Investigator, Shawn Leng-Hsien Soh, Principal Investigator, Queen Margaret University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REP 0197; 2019129 (Other: Singapore Institute of Technology)
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Accidental Fall; Aging; Self Efficacy

STUDY DESIGN:
Intervention Model Description: Phase 1 Participants will be requested to report the incidence of no fall, near-fall or a fall daily over the next 21-day period. There will be 3 options given to the participants: (1) a daily telephone call at a prearranged timing or (2) a daily text message given at a prearranged timing or both. A study administrator will contact the participant daily using the preferred mode of reporting. All information will be recorded in a logbook.
  Phase 2 The development of the Balance Recovery Falls-Efficacy scale will be guided using the COSMIN methodology. This development is based on inputs from the community-dwelling older adults to ensure relevance, comprehensiveness and comprehensibility. The scale would then be validated with a group of healthcare professionals and another new group of community-dwelling older adults using the Delphi method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Developing the list of items for BRFES (Experimental): Two groups of six community-dwelling older adults will participate in a focus group session. Each focus group session will begin with a trained facilitator using a session guide welcoming the participants and introducing the participants in the group. The session will adopt a nominal group method which includes silent generation of ideas, sharing of an idea in a 'round robin' fashion, group discussion to clarify ideas and then completing the session with anonymous voting to include items into a list of items to be included in the Balance Recovery Falls-Efficacy Scale (BRFES).
  Interventions: Other: Developing the list of items for BRFES

INTERVENTIONS:
Other: Developing the list of items for BRFES — The finalized list of items will be discussed by two researchers who will combine similar items generated by the two focus groups to complete the Balance Recovery Falls-Efficacy Scale. The list of items has been developed by a group of community-dwelling older adults who had demonstrated an understanding of near-falls and will be able to articulate the use of balance recovery strategies used in near-fall experiences.

SUMMARY:
The first phase of the study aims to study the incidence of near-falls. The second phase will be to develop a scale which operationalize balance recovery confidence in the older adults. This study will determine the incidence of near-falls in a sample of community-dwelling older adults and will develop the Balance Recovery Falls-Efficacy scale (BRFES) for the community-dwelling older adults using the COSMIN method. This scale will be used to measure the confidence level of the community-dwelling older adults in their ability to execute balance recovery maneuvers in common, everyday functional activities to prevent a fall.

DETAILED DESCRIPTION:
This study will progress through two phases

The first phase will recruit 30 older adults from ages of 65 and older living in the community. A study administrator will contact the participants daily over a 21-day period to obtain frequency and type of event experienced e.g. no fall, fall, near fall (hand), near-fall (leg) or near-fall (other). No other details of the event will be ascertained because this preliminary study will be to determine the incidence of near-falls in a sample of community-dwelling seniors.

The second phase will be to develop a scale which operationalize balance recovery confidence in community-dwelling older adults. In the first stage of the study, twelve older adults will be recruited to develop a comprehensive list of relevant items for the scale. Purposive sampling will be used to invite participants from the earlier study. This approach will ensure sample representativeness of the population and to include participants who have had demonstrated an understanding of near-falls and balance recovery maneuvres in the previous study to develop the scale. An exhaustive list of scale items will be generated from two focus group formed by six participants using a nominal group technique. This consensus-based technique ensures that all items in the scale are relevant and comprehensible to the community-dwelling older adults to discriminate the confidence level in one's ability to perform balance recovery maneuvres. The scale will then be sent to a panel of 50 experts including healthcare professionals as well as a new group of community-dwelling older adults to determine the appropriateness of items ensuring that the scale is relevant, comprehensive and comprehensible. Delphi technique will be adopted as the method to obtain a consensus among experts to finalize the Balance Recovery Falls-Efficacy Scale (BRFES).

ELIGIBILITY:
Inclusion Criteria:

* 65-year-old and above
* Ability to read, write and communicate in English
* History of at least one near-fall or one fall within the last 12 months
* Living independently in the community with or without the use of a walking aid
* Not having any cognitive dysfunction by achieving a score of 7 or less in the 6-item cognitive impairment test (6CIT)
* Able to walk 6 meters within 12 seconds by performing the Timed Up and Go (TUG) test
* Able to catch a 30cm ruler by each hands using the ruler drop test

Exclusion Criteria:

* Requiring any physical assistance from another person to walk within home
* Known active malignant conditions
* Cardiovascular conditions e.g. neurally mediated syncope, cardiac syncope, structural heart diseases e.g. aortic stenosis or hospitalization for myocardial infarction or heart surgery within 3 months
* Pulmonary conditions e.g. serious chronic obstructive pulmonary disease or oxygen dependence
* Musculoskeletal conditions e.g. moderate to severe osteoarthritis that could affect balance control and muscle function e.g. self-reported pain or dysfunction of the trunk and extremities, fractures or injuries in the extremities in the last 6 months
* Neurological conditions such as Parkinson's Disease, sequelae of stroke, Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS) or severe Dementia or epilepsy
* Legal blindness, severe visual impairment, severe hearing impairment or legal deafness

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of near-falls | 6 months
  To determine the incidence of near-falls
Development of the Balance Recovery Falls-Efficacy Scale (BRFES) | 9 months
  To develop and validate the Balance Recovery Falls-Efficacy Scale (BRFES).
  The construct measured is the confidence in one's ability to execute balance recovery manoeuvres in common, everyday functional activities to prevent a fall. The scale response option ranged from 1 to 10 with a higher score reflecting higher confidence. The scale would have 16 items indicating a total score range of 16 to 160. A higher total score value represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Soh, Principal Investigator — Singapore Institute of Technology
Locations (1):
- Singapore Institute of Technology, Singapore, Singapore

REFERENCES:
- [Derived] Soh SL, Tan CW, Lane J, Yeh TT, Soon B. Near-falls in Singapore community-dwelling older adults: a feasibility study. Pilot Feasibility Stud. 2021 Jan 12;7(1):25. doi: 10.1186/s40814-020-00748-1. PMID 33436025